CLINICAL TRIAL: NCT00341211
Title: Specimens From Normal Controls
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999996013; OH96-C-N013
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2010-12-01

CONDITIONS: Viral Infections
Keywords: AIDS; Cancer; Epidemiology; Immunology; Virology
MeSH Terms: conditions — Virus Diseases; Acquired Immunodeficiency Syndrome; Neoplasms

SUMMARY:
The Viral Epidemiology Branch (VEB) of the National Cancer Institute (NCI) conducts research on viral infections and their associations with various diseases including AIDS and cancer. For some research questions, specimens are available from "case" subjects as part of ongoing protocols but are not available from normal "control" subjects (i.e., those without the infection or disease under study) to whom the case subjects can be compared. This protocol is to obtain routine specimens (usually peripheral venous blood, occasionally other body fluid such as saliva, urine, or tears) from healthy volunteers.

DETAILED DESCRIPTION:
The Viral Epidemiology Branch (VEB) of the National Cancer Institute (NCI) conducts research on viral infections and their associations with various diseases including AIDS and cancer. For some research questions, specimens are available from "case" subjects as part of ongoing protocols but are not available from normal "control" subjects (i.e., those without the infection or disease under study) to whom the case subjects can be compared. This protocol is to obtain routine specimens (usually peripheral venous blood, occasionally other body fluid such as saliva, urine, or tears) from healthy volunteers.

ELIGIBILITY:
* INCLUSION CRITERIA:

Subjects can be friends of VEB investigator or collaborator, hospital or office workers, repeat volunteer blood donors, etc.

EXCLUSION CRITERIA:

Must not be minors, prisoners, pregnant women or incapable of providing informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 1996-04-11; Study Completion 2010-12-01

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Institute (NCI), 9000 Rockville Pike, Bethesda, Maryland, United States